CLINICAL TRIAL: NCT05956392
Title: Reducing Children's Screen Use for Better Sleep, Mental, and Brain Health: a Personalised Approach
Brief Title: Personalising Children's Screen Use Reduction for Better Sleep, Mental, and Brain Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, June Chi Yan Lo, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MEDRES
Record Dates: First submitted 2023-07-04; First posted 2023-07-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Screen-use Reduction + Sleep Extension; Free-living
Keywords: Cognitive Functions; Neurobehavioural Functions; Sleep Duration; Screen-use; High-density EEG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screen-use reduction + Sleep extension (Experimental): For the intervention group, participants are required to follow an agreed schedule where one hour of their daily screen-use time during school days will be repurposed for additional sleep during the two-week manipulation period.
  Interventions: Behavioral: Screen-use reduction + Sleep extension
- Free-living control (No Intervention): For the control group, participants will remain under free-living conditions (no restrictions on their screen-use time or sleep time) during the two weeks.

INTERVENTIONS:
Behavioral: Screen-use reduction + Sleep extension — 60 minutes of a participants' daily screen-use time on school days will be repurposed for more sleep time.
  Arms: Screen-use reduction + Sleep extension

SUMMARY:
In Singapore, 64.4% of school-age children sleep less than the minimum recommended duration of 9 hours on school nights, thus risking poor mental, cognitive, and brain health. These short-sleeping children, however, spend on average 2.5 hours per school day on non-academic media use, revealing the potential of reducing their screen time for more sleep. Previous interventions targeted at reducing media use and/or improving sleep among school-age children, though effective in increasing sleep, required cooperation from schools, extensive personnel training, and high commitment of participants, rendering them difficult to implement in Singapore. Existing interventions also focused on evening or pre-bedtime screen use, and took a one-size-fits-all approach, ignoring individual differences in the duration, type, and purpose of media use throughout the day. Here, we propose a scalable approach to curtail media use based on individual need throughout the day. We will conduct a randomised controlled trial during term time, recruiting 150 children, aged 6-12 years, who on school days, sleep less than 8 hours and spend more than 2 hours on media use. At baseline, all participants will record their time use patterns. The research staff will then help the intervention group to repurpose at least 60 minutes of media use per school day for sleep. Importantly, participants can decide the type, timing and duration of media use to curtail, thus giving them a sense of agency and mastery, while boosting their self-efficacy, a vital ingredient in behavioural change. The intervention group will follow this personalised schedule for 2 weeks, while the control group will be in a free-living condition. Two weeks after the intervention has ended, the intervention group will undergo follow-up assessments. Throughout the study, sleep, time use, cognitive functions, and psychological well-being will be assessed daily. Other cognitive tasks and questionnaires will be conducted during 2-3 lab/school-classroom visits, with one-third of the participants also undergoing high-density electroencephalography to measure brain activity.

DETAILED DESCRIPTION:
Design:

This study will be a randomised controlled trial that assesses the effectiveness of a personalised media use intervention on improving sleep, mood and cognitive functioning in school-aged children. The study will be conducted during term time. A total of 150 children aged from 6 to 12 years old will be recruited in Singapore. Participants will be randomly assigned to either an intervention or a control group.

Recruitment and screening:

Participants will be recruited via primary schools in Singapore, email lists, social media platforms (e.g. Facebook parent groups), flyers in the community and word-of-mouth.

In order to screen for eligibility, parents of interested participants will be invited to complete a screening questionnaire. This questionnaire will take approximately 5-10 minutes to complete. If at screening, they fulfill all the criteria for inclusion in the study, they will be invited to participate in the study. Inclusion in the study will be based on whether (1) The parent is between 25 and 60 years old, (2) The child is between 6 and 12 years old, (3) Both parent and child must be English speaking, (4) Child should be healthy (no sleep disorder, chronic illness, developmental condition, and should not be on any long-term medication), (5) both parent and child should either be a Singaporean Citizen or Permanent Residents, (6) child habitually sleeps < 8 h on school nights and should spend > 2 h on media use (i.e. social media, gaming, and TV / videos) on school days.

Briefing Session (Via video-call):

Venue: Through video-call Duration: ~30 minutes

A member of the research team will explain to the participant and their parent the aims and the procedures of the study. The participant and their parent will be provided with time for questions. If the participant and their parent agree to take part in the study, they will be asked to provide their written informed consent /assent several days before the start of the study. Teachers of the child will also undergo a similar briefing and consent taking procedure, but on a separate video-call.

Procedure:

The study protocol can be broken down into three periods - baseline, manipulation and follow-up period.

1) Baseline period

Venue: Participants' home and school Duration: 1 week

Participants from both intervention and control groups will be monitored under free-living conditions for 1 week to establish their regular sleep and daytime schedule. Their sleep at home will be objectively measured using actigraphy, as well as Fitbit devices which would allow for remote monitoring. The parent will be given a sleep diary which consists of an actiwatch removal log and a log for reporting details of the child's daytime nap and nocturnal sleep on a daily basis during participation in the study. Ecological momentary assessments (EMA) will be administered over a mobile phone loaned to participants and an application that was developed in-house will be used to assess participants' mood, sleepiness and cognitive functions on a daily basis.

The EMA tasks will take approximately 10 minutes per day and will include:

1. Karolinska Sleepiness Scale (10 seconds)
2. Positive and Negative Affect Schedule for Children (PANAS-C) for mood assessment
3. A Dot Memory Task which is a spatial working memory task requiring participants to remember and recall locations of dots placed on a 5x5 grid.
4. A Symbol Search Task that requires participants to match pairs of symbols displayed on the screen to measure their processing speed.
5. A 3-min Psychomotor Vigilance Task which is a simple reaction time task that will measure their sustained attention.

   Parents/caregivers will be asked to report their children's daily time use on a separate mobile phone application installed on their own phone. Parents/caregivers will log the child's daily activities at a 15-minute resolution by choosing from a list of primary activities customized for the current project (e.g. school, homework, travel, electronic device). Hardcopies of a time-use diary will be provided to caregivers who are not familiar with the mobile technology.

   On the last day of the baseline week, participants and their parent will be invited to the lab/school-classroom within the school compound for additional baseline assessments after school. In cases where parents are unable to make it to a face to face session at the lab/school-classroom, online sessions will be facilitated by our team to brief parents on how to complete these baseline assessments remotely.

   During the visit, participants will be required to complete the following questionnaires and tasks. A study team member will be present to verbally explain any questions/tasks that child participants are unable to understand. Participants will be allocated separate spaces to complete these tasks/questionnaires:

   1) Karolinska Sleepiness Scale (10 seconds) 2) A 10-min Psychomotor Vigilance Task that measures sustained attention. (10 mins) 3) 1-back and 2-back tasks that measure working memory/executive functions. Participants will be required to determine whether the alphabet currently shown on the computer screen is the same as the alphabet shown 1 or 2 items ago. (8 mins) 4) Symbol Digit Modalities Test which is a 2-minute task which measures speed of processing/cognitive throughput and requires participants to input a digit corresponding to the symbol shown based on a key provided. (2 mins) 5) Positive and Negative Affect Schedule for Children (PANAS-C) for mood assessment (10-mins) 5) Digital Addiction Scale for Children (DASC) that assesses digital device usage (5 mins)

   Parents/caregivers of participants are required to complete the following tasks through an online link which will be sent to them. Parents/caregivers are required to complete the following questionnaires over the Qualtrics platform:
   1. Parent-child Internet Addiction Test (PC-IAT) that measures the internet addiction symptoms(10 mins)
   2. Pediatric Daytime Sleepiness Scale (PDSS) that measures the child's sleepiness level (1 min)
   3. Child Behavioural Checklist-parent version (CBCL-P) that assesses the child's internalizing and externalizing behaviours (15 mins)
   4. Singapore Children Sleep Survey which is a questionnaire that assess children sleep behaviour and related factors (30-40 mins)

   Additionally, questionnaires will be sent via online links to the participant's teachers after the first week of the baseline period. Teachers of the participants are required to complete the following questionnaires over the Qualtrics platform:
   1. Child Behavioural Checklist- teacher version (CBCL-T) (15 mins)
   2. Karolinska Sleepiness Scale (10 seconds)

   For the intervention group, a research staff will also evaluate the time-use data collected from the first week with the child and parents and help them restructure their daily schedule during the baseline lab/school-classroom visit. In cases where parents are unable to make it to a face to face session at the lab/school-classroom, online sessions will be facilitated by our team to help them restructure their daily schedule.

   Participants are required to identify a minimum of 60 minutes spent on media use on each school day, which they will be willing to forego for more sleep during the subsequent manipulation period. Participants can decide the time of the day and duration of the type of media use that they would like to curtail in order to advance their bedtime.

   For the control group, participants will undergo the same cognitive tasks and complete the mood questionnaires as the intervention group. Parents/caregivers and teachers of participants will also be asked to complete the same battery of questionnaires on their children/students' behaviours and daytime sleepiness. However, participants will not be guided through a personalised schedule restructuring, and will remain under free-living conditions for the next two weeks.

   The lab/school-classroom visit is expected to last between 1 - 1.5 hours. If parents are unable to come in to the lab/school-classroom for the first visit, the online 1 on 1 session will also be expected to last between 1-1.5 hours.

   2) Manipulation period

   Venue: Participants' home and lab/school-classroom Duration: 2 weeks

   For the intervention group, participants are required to follow the agreed schedule to reduce their media use during the two-week manipulation period. Sleep measurement and EMA will be performed in the same manner as they were during the baseline period. Parents/caregivers and teachers will be asked to complete the same tasks/questionnaires as at the first lab/school-classroom visit. In cases where parents are unable to make it to a face to face session at the lab/school-classroom, online sessions will be facilitated by our team to help them complete these tasks/questionnaires remotely. After the first week of the manipulation period, research staff will schedule an online session to resolve any problems in following the new schedules. Research staff will closely monitor the participants' sleep and media use using the Fitbit devices as well as the online time use app to ensure the correct usage and compliance with the new schedule. Research staffs will contact and help participants in case of any observed deviations.

   For the control group, participants will complete the same sleep assessments and EMA as during the baseline period, and will remain under free-living conditions during the two weeks.

   After two weeks of manipulation, participants will be invited back to the lab/school-classroom to undergo the same cognitive assessments and questionnaires as the first lab/school-classroom visit.

   For the intervention group, participants will also report their level of satisfaction with the new sleep schedule and time use and indicate the likelihood of continuing with the tailored-made schedule in the future.

   For the control group, a one-to-one consultation will be conducted by a research staff who will help then re-allocate at least 60 min of their media use time for sleep. Thus, even the control group can benefit from the intervention. This lab/school-classroom visit will be the last session for participants in the control group. In cases where participant's parents are unable to make it to a face to face session at the school-classroom, online sessions will be facilitated by our team to help the parent-child dyad restructure their daily schedule.

   3) Follow-up period

   Venue: Participants' home and school-classroom/laboratory Duration: 1 week

   Participants in the intervention group will be invited to complete the same questionnaires and tasks using actigraphy and Fitbit as well as the EMA and time-use applications over a 1-week follow-up period. Participants will also be asked to fill in sleep diaries on a daily basis. This follow-up period will take place two weeks after the end of the manipulation period.

   Upon the completion of the follow-up period, participants will be invited for their final lab/school-classroom visit where they will be asked to undergo the same procedure as the previous lab/school-classroom visits (baseline visit) for the assessment of mood, sleepiness, device use and cognitive functioning.

   Parents/caregivers and teachers will be asked to complete the same questionnaires as given during the previous(baseline and manipulation) lab/school-classroom visits. In cases where parents are unable to make it to a face to face session at the lab/school-classroom, online sessions will be facilitated by our team to brief parents on how to complete these assessments remotely.

   If child participants are undergoing study procedures at the NUS laboratory, parents will still have to attend the session face-to-face with their child.

   High-density EEG measures For both the intervention group and the control group, a subset of the participants (n= 20 for each group) will undergo the high-density EEG during lab visits (i.e. 3 times for the intervention group and twice for the control group). EEG data will be measured for 5 minutes of resting state and the EEG power and coherence of the prefrontal cortex will be studied. Research has shown that the brain activity in the prefrontal cortex is associated with the attention network and its function. The natural-logged ratio of theta/beta power for frontal leads will be used in the subsequent analyses.

ELIGIBILITY:
Inclusion Criteria:

* Is a Singaporean or Permanent Resident
* Speaks English
* Aged between 6-12 years old
* Habitually sleeps less than 8 hours during school nights
* Habitually spends more than 2 hours on media use (i.e. social media, gaming, and TV / videos) on school days
* Is not on any long-term medications
* Has no known medical or developmental conditions that could affect sleep (e.g. asthma, arthritis, cancer, congenital heart disease, diabetes, epilepsy, eczema, inflammation)
* Has no history of psychiatric or neurological disorders

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sustained attention assessed with the Psychomotor Vigilance Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PVT will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again at the end of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Number of attention lapses. More lapses indicate worse performance.
Change in sustained attention assessed with the Psychomotor Vigilance Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PVT will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again at the end of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Mean reaction time. Longer mean reaction time indicate worse performance.
Change in sustained attention assessed with the Psychomotor Vigilance Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PVT will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again at the end of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Median reaction time. Longer median reaction time indicate worse performance.
Change in sustained attention assessed with the Psychomotor Vigilance Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PVT will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again at the end of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Standard deviation in reaction time. Larger standard deviation in reaction time indicate less consistent performance.
Change in sustained attention assessed with the Psychomotor Vigilance Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PVT will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again at the end of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Number of commission errors/false starts. More false starts indicate worse performance.
Change in number of correct matches assessed with the 1-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of correct matches in the 1-back task. More correct matches indicate better performance.
Change in number of incorrect matches assessed with the 1-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of incorrect matches in the 1-back task. Fewer incorrect matches indicate better performance.
Change in number of correct mismatches assessed with the 1-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of correct mismatches in the 1-back task. More correct mismatches indicate better performance.
Change in number of incorrect mismatches assessed with the 1-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of incorrect mismatches in the 1-back task. Fewer incorrect mismatches indicate better performance.
Change in discriminability measure (A') assessed with the 1-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Discriminability measure (A')
Change in bias measure (B"D) assessed with the 1-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | On the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Bias measure (B"D)
Change in number of correct matches assessed with the 2-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of correct matches in the 2-back task. More correct matches indicate better performance.
Change in number of incorrect matches assessed with the 2-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of incorrect matches in the 2-back task. Fewer incorrect matches indicate better performance.
Change in number of correct mismatches assessed with the 2-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of correct mismatches in the 2-back task. More correct mismatches indicate better performance.
Change in number of incorrect mismatches assessed with the 2-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of incorrect mismatches in the 2-back task. Fewer incorrect mismatches indicate better performance.
Change in discriminability measure (A') assessed with the 2-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Discriminability measure (A')
Change in bias measure (B"D) assessed with the 2-back task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Bias measure (B"D)
Change in subjective sleepiness assessed with the Karolinska Sleepiness Scale from baseline to manipulation (for both groups), baseline to follow-up (for intervention group only), and manipulation to follow-up period (for intervention group only) | KSS will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Score on the Karolinska Sleepiness Scale (1-9 points). Higher score indicate more sleepiness.
Change in positive mood from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PANAS-C will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Total score on the positive subscale of the Positive and Negative Affect Schedule for Children(PANAS-C) ranges between 5 and 25. A higher score indicates more positive mood and is considered to be better.
Change in negative mood from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | PANAS-C will be assessed once daily (up to 3 weeks for the control group and up to 4 weeks for the intervention group) using EMA, and again on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery.
  Total score on the negative subscale of the Positive and Negative Affect Schedule for Children(PANAS-C) ranges between 5 and 25. A higher score indicates more negative mood and is considered to be worse.
Change in processing speed assessed with the Symbol Digit Modalities Test from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Number of correct responses in the task
Change in digital device use assessed by the Digital Addiction Scale for Children from baseline to manipulation (for both groups), baseline to follow-up (for intervention group only), and manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  The Digital Addiction Scale for Children consists of 25 items rated on a five-point Likert scale ranging from 1 (Never) to 5 (Always). A total score is obtained by summing all 25 items (ranging from 25 to 125), with higher scores indicating a higher level of digital addiction.
Change in spatial working memory performance assessed by a Dot Memory Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Assessed once daily using EMA in both the control (up to 3 weeks) and intervention (up to 4 weeks) groups. The specific time at which the EMA is attempted daily (within a one hour time frame) is decided based on the participant's choice.
  Number of correct responses in the task. More correct responses indicate better performance.
Change in speed of processing assessed with a Symbol Search Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Assessed once daily using EMA in both the control (up to 3 weeks) and intervention (up to 4 weeks) groups. The specific time at which the EMA is attempted daily (within a one hour time frame) is decided based on the participant's choice.
  Number of correct responses in the task. More correct responses indicate better performance.
Change in speed of processing assessed with a Symbol Search Task from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Assessed once daily using EMA in both the control (up to 3 weeks) and intervention (up to 4 weeks) groups. The specific time at which the EMA is attempted daily (within a one hour time frame) is decided based on the participant's choice.
  Median reaction time. Longer median reaction time indicate worse performance.
Change in daily screen-use time assessed with time-use diary from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Assessed once daily using EMA in both the control (up to 3 weeks) and intervention (up to 4 weeks) groups. The specific time at which the EMA is attempted daily (within a one hour time frame) is decided based on the participant's choice.
  Time spent on electronic devices daily
Change in sleep duration from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Assessed daily using an actiwatch, fitbit and time-use app/sleep diary. Up to a total of 3 weeks in control participants and up to a total of 4 weeks of daily monitoring in intervention participants.
  Time spent sleeping will be assessed through an Actiwatch and the Fitbit worn by the children during the entire course of the study. The time-use app and the sleep diary filled in by parents daily during participation in the study will also help us gain a complete understanding of changes in sleep duration patterns throughout study participation.
Change in sleep efficiency from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Assessed daily using an actiwatch. Up to a total of 3 weeks in control participants and up to a total of 4 weeks of daily monitoring in intervention participants.
  Sleep efficiency will be assessed through an actiwatch worn throughout participation in the study.
Change in subjective sleepiness ratings by parents and teachers from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once one the last day of the baseline, manipulation and follow-up period through an online questionnaire sent to parents and teachers. Up to twice in the control group participants and up to thrice in intervention group participants.
  Subjective sleepiness will be assessed through the Pediatric Daytime Sleepiness Scale (PDSS) done by the child's parent and teacher. Score will range between 0 and 32 where higher scores indicate more sleepiness.
Change in subjective sleepiness ratings by parents and teachers from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once one the last day of the baseline, manipulation and follow-up period through an online questionnaire sent to parents and teachers. Up to twice in the control group participants and up to thrice in intervention group participants.
  Subjective sleepiness will also be assessed through the Karolinska Sleepiness Scale (KSS) done by parents and teachers. The KSS measures subjective sleepiness on a scale of 1='very alert' to 9='very sleepy, fighting sleep. Higher scores indicate more sleepiness.
Change in internet addiction symptoms from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Assessed using the Parent-child Internet Addiction Test (PC-IAT) which will indicate the level of problematic behaviour associated with compulsive use of electronic devices
Change in internalising and externalising behaviours from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Assessed using the Child Behavioural Checklist done by both parents and teachers.
Change in parent-reported sleep behaviours and sleep-related factors from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Assessed using the Singapore Children Sleep Survey done by parents.
Change in EEG power and coherence of the prefrontal cortex from baseline to manipulation (for both groups), from baseline to follow-up (for intervention group only), and from manipulation to follow-up period (for intervention group only) | Once on the last day of the baseline, manipulation and follow-up period through a laptop-based test battery. Up to twice in the control group and up to thrice in intervention group participants.
  Assessed using high-density EEG. he natural-logged ratio of theta/beta power for frontal leads will be used in the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: June Lo, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No